CLINICAL TRIAL: NCT01812837
Title: The Use of Microneedles in Photodynamic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 282150
Record Dates: First submitted 2013-03-13; First posted 2013-03-18 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; microneedles; photodynamic therapy; levulan; Aminolevulinic acid
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Blue Light

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 20 minutes incubation - with pretreatment (Experimental)
  Interventions: Device: Microneedle; Drug: Aminolevulinic Acid; Radiation: Blue light
- 40 minutes incubation - with pretreatment (Experimental)
  Interventions: Device: Microneedle; Drug: Aminolevulinic Acid; Radiation: Blue light
- 60 minutes incubation - with pretreatment (Experimental)
  Interventions: Device: Microneedle; Drug: Aminolevulinic Acid; Radiation: Blue light
- 60 minutes incubation - no pretreatment (Sham Comparator)
  Interventions: Drug: Aminolevulinic Acid; Radiation: Blue light

INTERVENTIONS:
Device: Microneedle — The study device (Microchannel Skin System by 3M Company)is fabricated from medicalgrade polymer consisting of a rectangular array of 351 pyramidal, 700-μm-long, solid microneedles.
  Other Names: Microchannles
  Arms: 20 minutes incubation - with pretreatment; 40 minutes incubation - with pretreatment; 60 minutes incubation - with pretreatment
Drug: Aminolevulinic Acid — Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
Radiation: Blue light — Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA)

SUMMARY:
The global aim of this study is to investigate how microneedles can facilitate the penetration and efficacy of photodynamic therapy in the treatment of actinic keratoses

The specific aims are as follows:

1. Investigate whether pretreatment with microneedles enhances penetration of topical aminolevulinic acid (ALA) that is marketed as Levulan® Kerasticks by DUSA pharmaceuticals Inc.
2. Investigate whether pretreatment with microneedles can decrease the required incubation times of the topical ALA prior to exposure to blue light photodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are 18 and older
2. Subjects who have at least 3 actinic keratoses on each side of the forehead
3. Subjects who signed an IRB approved informed consent

Exclusion Criteria:

1. Subjects who smoke
2. Subjects who have a photosensitizing condition such as lupus, porphyria, or similar condition.
3. Subjects who received a diagnosis of skin cancer on the face in past year
4. Subjects who received field treatment for actinic keratoses to the face in the past 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis, Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical

RESULTS

PARTICIPANT FLOW:
Groups:
- 20 Minute Microneedle Pretreatment Incubation: 20 min microneedle pretreatment incubation vs standard 60 min incubation (split-face)
  Microneedle: The study device (Microchannel Skin System by 3M Company)is fabricated from medicalgrade polymer consisting of a rectangular array of 351 pyramidal, 700-μm-long, solid microneedles.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA)
- 40 Minute Microneedle Pretreatment Incubation: 40 min microneedle pretreatment incubation vs standard 60 min incubation (split-face)
  Microneedle: The study device (Microchannel Skin System by 3M Company)is fabricated from medicalgrade polymer consisting of a rectangular array of 351 pyramidal, 700-μm-long, solid microneedles.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA)
- 60 Minute Microneedle Pretreatment Incubation: 60 min microneedle pretreatment incubation vs standard 60 min incubation (split-face)
  Microneedle: The study device (Microchannel Skin System by 3M Company)is fabricated from medicalgrade polymer consisting of a rectangular array of 351 pyramidal, 700-μm-long, solid microneedles.
  Aminolevulinic Acid: Levulan® Kerastick® DUSA Pharmaceuticals, Inc., Wilmington, MA
  Blue light: Blu-U unit (DUSA Pharmaceuticals, Inc., Wilmington, MA)
Period: Overall Study
Arm/Group | 20 Minute Microneedle Pretreatment Incubation | 40 Minute Microneedle Pretreatment Incubation | 60 Minute Microneedle Pretreatment Incubation
Started | 17 | 17 | 17
Completed | 15 | 16 | 17
Not Completed | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 Minute Microneedle Pretreatment Incubation | 40 Minute Microneedle Pretreatment Incubation | 60 Minute Microneedle Pretreatment Incubation | Total
Number analyzed (Participants) | 17 | 17 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 9 | 21
  >=65 years | 13 | 9 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (6.4) | 66.9 (9.8) | 66.2 (10.3) | 67.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 8
  Male | 14 | 16 | 13 | 43
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Actinic Keratoses Reduction Percent
Time Frame: one month after treatment
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 20 Minute Microneedle Pretreatment Incubation | 40 Minute Microneedle Pretreatment Incubation | 60 Minute Microneedle Pretreatment Incubation
Number analyzed (Participants) | 15 | 16 | 17
percentage
  Microneedle Pretreatment | 71.4 (22.6) | 80.2 (18.7) | 72.5 (22.8)
  Control | 68.3 (13.0) | 80.1 (18.1) | 73.6 (28.3)

ADVERSE EVENTS:
Arm/Group | 20 Minute Microneedle Pretreatment Incubation | 40 Minute Microneedle Pretreatment Incubation | 60 Minute Microneedle Pretreatment Incubation
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No